CLINICAL TRIAL: NCT05184374
Title: Efficacy of Prolonged Gonadorelin Stimulation Test in Male Adolescents With Postoperative Hypogonadotropic Hypogonadism
Brief Title: Efficacy of Prolonged GnRH Test in Male Adolescents With Postoperative HH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, vice director of endocrine department, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2021-674
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subcutaneous injection of gonadorelin is facilitated by GnRH pump (Experimental): After non-dose GnRH stimulation test on day 1, GnRH pump pulse subcutaneous injection of gonadorelin on the next day until one month.
  Interventions: Drug: Gonadorelin

INTERVENTIONS:
Drug: Gonadorelin — GnRH pump pulse subcutaneous injection of gonadorelin in a month

SUMMARY:
The Hypogonadotropic Hypogonadism(HH) could be caused by sellar lesions, sellar surgery or sellar radiotherapy. The incidence of HH after sellar surgery was higher in men than in women, and the therapy of HH was insufficient. Gonadotropin-releasing hormone(GnRH) stimulation test is used to evaluate the function of pituitary-gonadal axis. GnRH can be used to diagnose and treat fertility disorders and other endocrine disorders caused by HH. After a single injection of GnRH, the patients with poor response of luteinizing hormone and follicle stimulating hormone need to take extended provocation test, which is conducive to the formulation of the following treatment. GnRH pump can pulse subcutaneous injection of gonadorelin, which can be used as the extended provocation test.

ELIGIBILITY:
Inclusion Criteria:

* patients with HH after surgery of the saddle area
* sufficient therapy of the hypothalamic-pituitary-adrenal(HPA) and hypothalamic-pituitary-thyroid(HPT) axis

Exclusion Criteria:

* contradictions to gonadorelin
* androgen-dependent prostate cancer
* on the therapy of human chorionic gonadotropin(HCG) or testosterone

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — the changes of LH, FSH are complicated during the menstrual cycle, so female was excluded.
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
level of luteinizing hormone, follicle stimulating hormone and testosterone | 1 month
  after the GnRH pump of gonadorelin, the level of luteinizing hormone, follicle stimulating hormone and testosterone will be measured at 24h, 1, 2, 3 and 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China